CLINICAL TRIAL: NCT04528667
Title: A Phase 2, Randomized, Double-Blind, Placebo-controlled Study of the Safety and Efficacy of STI-5656 (Abivertinib Maleate) in Subjects Hospitalized Due to COVID-19
Brief Title: Study of the Safety and Efficacy of STI-5656 (Abivertinib Maleate) in Subjects Hospitalized Due to COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BTK-COV-202BR
Record Dates: First submitted 2020-08-20; First posted 2020-08-27 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Covid19
Keywords: covid-19
MeSH Terms: conditions — COVID-19 | interventions — abivertinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STI-5656 (Experimental): STI-5656 (abivertinib maleate) capsules administered orally 100 mg QD for 7 days, in addition to standard of care
  Interventions: Drug: STI-5656
- Placebo (Placebo Comparator): Placebo capsules administered orally daily for 7 days, in addition to standard of care
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: STI-5656 — STI-5656 (abivertinib maleate) is a third-generation EGFR tyrosine kinase inhibitor and BTK Inhibitor.
  Other Names: abivertinib maleate; avitinib; AC0010; abivertinib
  Arms: STI-5656
Drug: Placebo — Placebo capsules
  Arms: Placebo

SUMMARY:
A phase 2, placebo-controlled study of the safety and efficacy of STI-5656 (Abivertinib Maleate) in subjects hospitalized due to COVID-19

DETAILED DESCRIPTION:
This is a phase 2, randomized, double-blind, placebo-controlled study of the safety and efficacy of STI-5656 (Abivertinib Maleate) in subjects hospitalized due to COVID-19 in Brazil. Subjects are randomized 3:1 STI-5656 to placebo. Subjects receive either 100 mg of STI-5656 or placebo daily for 7 days. Standard of care will be maintained for all subjects throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed positive for COVID-19 by RT-PCR assay or equivalent
* Subject or family member/caregiver must have provided written informed consent which includes signing the institutional review board (IRB) or independent ethics committee (IEC) approved consent form prior to participating in any study related activity. However, if obtaining written informed consent is not possible, other procedures as provided in the March 27, 2020 (Updated on July 2, 2020) FDA Guidance on Conduct of Clinical Trials of Medical Products during COVID-19 Pandemic, Question 10, may be used
* Able to swallow capsules
* Willing to follow contraception guidelines

Exclusion Criteria:

* Pregnant or breast feeding
* Suspected uncontrolled active bacterial, fungal, viral, or other infection other than COVID-19
* Treatment with a strong cytochrome p450 3A4 inhibitor or inducer within 7 days prior to Day 1
* Received anti-rejection or immunomodulatory drugs within 14 days prior to Day 1
* Concurrent participation in another clinical trial involving therapeutic interventions (observation studies are acceptable)
* Any condition that confounds the ability to interpret data from the study
* Any significant medical condition, laboratory abnormality, or psychiatric illness that would interfere with or prevent the subject from participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects discharged from hospital | Randomization through Day 29
  Proportion of subjects whoa re alive and discharged from the hospital by Day 29

SECONDARY OUTCOMES:
Incidence of adverse events (safety) | Randomization through study completion through Day 36
  Types, frequencies, and severities of adverse events and their relationships to STI-5656, including serious adverse events
Time to hospital admission, treatment, and discharge | Randomization through study completion through Day 36
  Time from onset of COVID-19 symptoms to hospital admission, time from hospitalization to start of treatment (D1), and time from D1 to hospital discharge
Number of days hospitalized | Randomization to Day 36
  Number of days hospitalized from randomization through Day 36
Change in clinical status as assessed using a 0-8 ordinal scale | Randomization to Day 3, Day 10, and Day 36
  Change in clinical status as assessed using a 0-8 ordinal scale, where a lower score equals better outcome, at Days 3, 10, and 36
Change in RT-PCR test results | Randomization to Day 3, Day 10, and Day 36
  Change in RT-PCR test results (or equivalent) at Days 3, 10, and 36
Change in C-reactive protein levels | Randomization to Day 3 and Day 10
  Change in C-reactive protein (CRP) levels at Day 3 and Day 10
AUC of STI-5656 (PK) | Randomization through Day 8
  Area under the serum concentration-time curve (AUC) of STI-5656
Cmax of STI-5656 (PK) | Randomization through Day 8
  Maximum observed serum concentration (Cmax) of STI-5656
t½ of STI-5656 (PK) | Randomization through Day 8
  Apparent serum terminal elimination half life (t½) of STI-5656
Change in cytokine levels | Randomization to Day 3 and Day 10
  Change in cytokine levels (including IL-6, TNF-a, IFNγ, IL1β) at Day 3 and Day 10
Tmax of STI-5656 (PK) | Randomization through Day 8
  Time to Cmax (Tmax) of STI-5656

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.
Locations (1):
- Hospital e Maternidade Christovão da Gama, Santo André, São Paulo, Brazil